CLINICAL TRIAL: NCT05520333
Title: Brief Intervention to Prevent Alcohol Socialization / Better Informed Parents Keeping Adolescents Safe From Alcohol (BIPAS Alcohol)
Brief Title: Brief Intervention to Prevent Alcohol Socialization (BIPAS Alcohol)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0101; 1R34AA028856-01A1 (NIH)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Drinking, Adolescent; Drinking Behavior; Drinking, Alcohol; Adolescent Behavior
MeSH Terms: conditions — Underage Drinking; Drinking Behavior; Alcohol Drinking; Adolescent Behavior | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Families receive text messages for three months.
  Interventions: Behavioral: BIPAS Alcohol
- Waitlist-control arm (No Intervention): Families are randomized into a control group for three months and begin receiving text messages for three months.

INTERVENTIONS:
Behavioral: BIPAS Alcohol — Weekly text messages for three months.
  Arms: Intervention arm

SUMMARY:
Early alcohol socialization occurs within the family. This multi-level, high-reach, low-intensity intervention to prevent early alcohol use capitalizes on the influence of providers, immunization timing, and pediatric guidelines that advise healthcare providers to give anticipatory guidance about early alcohol use. In conjunction, the intervention capitalizes on the power of technology to reinforce and expand upon pediatrician messages.

The study seeks to understand the feasibility and effectiveness of a pilot intervention designed to prevent alcohol socialization through education of parents of rising 6th grade students.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Parent or guardian of an enrolled child at a study clinic;
* Cohabitate part time (2 days/week) or more with enrolled child;
* Be able to complete study activities in English;
* Be able to give informed consent;
* Own a phone with text message capabilities and access to internet.

Exclusion Criteria:

* Families in which the 10-to-12-year old child is actively receiving treatment for alcohol use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilkey, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will be following NIAAA's requirements regarding sharing outcome data of sharing de-identified, individual-level data to the NIAAA Data Archive. The data are made public after an embargo period following the end date of the research award.
Time Frame: after an embargo period following the end date of the research award
Access Criteria: In accordance with NIAAA data archive requirements.
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from May to November 2023. Participants were recruited through school newsletters, social media posts, information dissemination through educational institutions and local pediatric clinics, and word of mouth.
Pre-assignment Details: Parent-child dyads participated in this study, but only parents/caregivers were considered enrolled. The number started/completed reflects the number of individual parents/caregivers.
Groups:
- Waitlist-control Arm: Families are randomized into a waitlist control group for three months and begin receiving text messages for three months.
Period: Overall Study
Arm/Group | Intervention Arm | Waitlist-control Arm
Started (The number started reflects the number of parents.) | 69 | 63
Completed | 66 | 57
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Population: Note that demographics were only collected for parent participants (not children).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Waitlist-control Arm | Total
Number analyzed (Participants) | 69 | 63 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 63 | 132
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study was not designed to collect these data; therefore, sex data were not collected.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 66 | 57 | 123
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 61 | 52 | 113
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 4 | 5
Parent drinks alcohol [Count of Participants; unit: Participants]
  Yes | 56 | 47 | 103
  No | 13 | 16 | 29
Parent/guardian relationship with child [Count of Participants; unit: Participants] — Parents' self-identified relationship with their child.
  Participants
    Mother | 61 | 54 | 115
    Father | 8 | 8 | 16
    Guardian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Value of Parental Pro-sipping Beliefs Score
Description: Parental Alcohol Socialization Beliefs, Attitudes, and Practices scale (eight items). A four-point scale ranging from "strongly disagree" (lowest value=1) to "strongly agree" (highest value=4) will be used, with higher values on the scale indicating a more pro-sipping belief system. The scores will have a range from 8-32. Higher values are associated with worse outcomes.
Time Frame: Baseline, three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Waitlist-control Arm
Number analyzed (Participants) | 66 | 57
score on a scale | 0.13 (0.14) | 0.08 (0.16)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse events data was not collected as part of this protocol.
Arm/Group | Intervention Arm | Waitlist-control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT05520333/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT05520333/ICF_000.pdf